CLINICAL TRIAL: NCT03463902
Title: Transcranial Direct Current Stimulation (tDCS) to Improve Gesture Control in Schizophrenia - a Randomised, Placebo-controlled, Double-blind Crossover Trial
Brief Title: Transcranial Direct Current Stimulation (tDCS) to Improve Gesture Control
Acronym: GesttDCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment failed to enroll sufficient number of patients
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-01995
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Gesture; tDCS; schizophrenia; nonverbal communication
MeSH Terms: conditions — Schizophrenia; Gestures; Nonverbal Communication

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, cross-over trial of 5 tDCS protocols
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: participants, outcome assessors and raters are blinded. tDCS application is performed by an unblinded investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- left IFG anodal (Experimental): 2 mA Stimulation of 10 min, anodal electrode over left IFG, cathodal electrode over right IFG, 30 sec ramp to start and 30 sec ramp to stop
  Interventions: Device: left IFG anodal
- left IFG cathodal (Active Comparator): 2 mA Stimulation of 10 min, cathodal electrode over left IFG, anodal electrode over right IFG, 30 sec ramp to start and 30 sec ramp to stop
  Interventions: Device: left IFG cathodal
- left IPL anodal (Active Comparator): 2 mA Stimulation of 10 min, anodal electrode over left IPL, cathodal electrode over right IPL, 30 sec ramp to start and 30 sec ramp to stop
  Interventions: Device: left IPL anodal
- left IPL cathodal (Active Comparator): 2 mA Stimulation of 10 min, anodal electrode over left IFG, cathodal electrode over right IFG, 30 sec ramp to start and 30 sec ramp to stop
  Interventions: Device: left IPL cathodal
- Placebo (Placebo Comparator): anodal electrode over left IFG, cathodal electrode over right IFG, stimulation only during 30 sec ramp at beginning and end of 10 min
  Interventions: Device: Placebo

INTERVENTIONS:
Device: left IFG anodal — Single session of transcranial direct current stimulation (tDCS) over left IFG anodal stimulation
  2 mA Stimulation of 10 min, anodal electrode over left IFG, cathodal electrode over right IFG, 30 sec ramp to start and 30 sec ramp to stop
  Arms: left IFG anodal
Device: left IFG cathodal — Single session of transcranial direct current stimulation (tDCS) over left IFG cathodal stimulation
  2 mA Stimulation of 10 min, cathodal electrode over left IFG, anodal electrode over right IFG, 30 sec ramp to start and 30 sec ramp to stop
  Arms: left IFG cathodal
Device: left IPL anodal — Single session of transcranial direct current stimulation (tDCS) over left IPL anodal stimulation 2 mA Stimulation of 10 min, anodal electrode over left IPL, cathodal electrode over right IPL, 30 sec ramp to start and 30 sec ramp to stop
  Arms: left IPL anodal
Device: left IPL cathodal — Single session of transcranial direct current stimulation (tDCS) over left IPL cathodal stimulation 2 mA Stimulation of 10 min, anodal electrode over left IFG, cathodal electrode over right IFG, 30 sec ramp to start and 30 sec ramp to stop
  Arms: left IPL cathodal
Device: Placebo — Single session of placebo tDCS over left IFG 10 min duration, 30 sec ramp during start and end
  Arms: Placebo

SUMMARY:
The majority of schizophrenia patients is impaired in hand gesture performance, which contributes to poor functional outcome and poor communication skills. The left inferior frontal gyrus (IFG) and the left inferior parietal lobe (IPL) are key nodes of the gesture network, which is less active in patients with schizophrenia. Here, the investigators test single 10 min sessions of tDCS known to either enhance or inhibit local brain activity for app. 1 hour. The investigators aim to determine, which protocol may improve gesture performance in patients and healthy controls. This is a randomized, double-blind, cross-over, placebo-controlled single-center trial in 20 patients with schizophrenia spectrum disorders and 20 healthy controls. Gesture performance will be tested immediately after each tDCS session, which are separated by 24 hours. Results of this study will inform larger interventional trials comparing 2 tDCS protocols with repeated administration.

DETAILED DESCRIPTION:
Schizophrenia is associated with poor social functioning, which is perturbed by deficits in social interaction including nonverbal communication. The use of hand gestures is critical for nonverbal communication, but the majority of schizophrenia patients has severe gesture impairments. Today no intervention may ameliorate gesture impairments.

Patients with gesture impairments have altered structure and function of the gesture network, particularly the left inferior frontal gyrus (IFG) and also the left inferior parietal lobe (IPL). Noninvasive brain stimulation techniques may alter local brain function. Transcranial direct current stimulation (tDCS) for 10 mins is a very safe method to alter brain states locally for a period of 1-2 hours. Indeed, facilitatory stimulation of the left frontal cortex by tDCS demonstrated improved gesture perception and interpretation in healthy subjects. Furthermore, patients with apraxia identified gestures better after facilitatory tDCS over the left inferior parietal lobe (IPL). Thus, the investigators hypothesize that local changes of brain activity within the gesture network would change gesture performance.Particularly, anodal (facilitatory) stimulation of the left IFG would improve gesture performance. The investigators will test single sessions of tDCS in healthy subjects and schizophrenia patients. If one of the protocols proves to have superior effects, this result will help to plan interventional trials targeting social interaction deficits in schizophrenia.

The aim of the study is to determine the effect of one 10 min session of anodal tDCS over the left IFG on gesture performance compared to three active and one placebo tDCS sessions. This is a randomized, double-blind, cross-over, placebo-controlled single-center trial in 20 patients with schizophrenia spectrum disorders and 20 healthy controls. After baseline assessment of gesture performance, participants will receive one 10 min tDCS protocol each day, immediately followed by assessments of gesture performance and dexterity. Gesture performance will be measured with video recorded Test of Upper Limb Apraxia, which is rated blindly according to a manual. Active comparisons are cathodal tDCS over left IFG, anodal tDCS over left IPL and cathodal tDCS over left IPL.

ELIGIBILITY:
Inclusion Criteria:

* Right handed according to the Edinburgh Handedness Inventory
* Ability and willingness to participate in the study
* Ability to provide written informed consent
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Spent majority of childhood/adolescence in Switzerland
* Patients: schizophrenia spectrum disorder according to DSM-5

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Metal objects on or in the body (e.g. grenade splinter, cardiac pacemaker, vessel clips, metal prostheses, contraceptive coil, cochlear implants, hearing aid, tooth implant)
* Tattoos on head, neck or shoulder in close proximity to the electrode placement
* Current skin problems on the scalp, eg. bruises or open wounds
* History of neurosurgery, any severe head wounds, history of neurologic disorders impacting gesture, e.g. Parkinson's disease, stroke, multiple sclerosis
* Active drug addiction except nicotine
* Known contact allergies
* Controls: first-degree relatives with schizophrenia spectrum disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Test of Upper Limb Apraxia | 10 mins after baseline assessment
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment and group
Test of Upper Limb Apraxia | 10 mins after tDCS intervention left IFG anodal
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment and group
Test of Upper Limb Apraxia | 10 mins after tDCS intervention left IFG cathodal
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment and group
Test of Upper Limb Apraxia | 10 mins after tDCS intervention left IPL anodal
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment and group
Test of Upper Limb Apraxia | 10 mins after tDCS intervention left IPL cathodal
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment and group
Test of Upper Limb Apraxia | 10 mins after tDCS intervention with placebo
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment and group

SECONDARY OUTCOMES:
Coin Rotation | 20 mins after baseline assessment
  Test of dexterity, 3 trials of 10s to rotate a .5 SFr coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns
Coin Rotation | 20 mins after tDCS intervention left IFG anodal
  Test of dexterity, 3 trials of 10s to rotate a .5 SFr coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns
Coin Rotation | 20 mins after tDCS intervention left IFG cathodal
  Test of dexterity, 3 trials of 10s to rotate a .5 SFr coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns
Coin Rotation | 20 mins after tDCS intervention left IPL anodal
  Test of dexterity, 3 trials of 10s to rotate a .5 SFr coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns
Coin Rotation | 20 mins after tDCS intervention left IPL cathodal
  Test of dexterity, 3 trials of 10s to rotate a .5 SFr coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns
Coin Rotation | 20 mins after tDCS intervention with placebo
  Test of dexterity, 3 trials of 10s to rotate a .5 SFr coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Walther, MD, Principal Investigator — University of Bern, University Hospital of Psychiatry
Locations (1):
- University Hospital of Psychiatry, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share the data, because they cannot anonymize the video data sufficiently